CLINICAL TRIAL: NCT01019330
Title: Radial Versus Femoral Arterial Access for Cardiac Catheterization: Comparison of Complications at 30 Days
Status: Completed | Type: Observational
Sponsor: Creighton University (Other)
Responsible Party: Sponsor
Other Study IDs: 09-15552
Record Dates: First submitted 2009-11-20; First posted 2009-11-25 (Estimated); Last update posted 2015-11-30 (Estimated); Status verified 2015-11

CONDITIONS: Radial Artery Occlusion
Keywords: radial vs femoral; radial artery cardiac catheterization
MeSH Terms: conditions — Arterial Occlusive Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Femoral: Subjects receiving femoral artery cardiac catheterization
  Interventions: Other: Distal pulses
- Radial: Subjects receiving radial artery cardiac catheterization
  Interventions: Other: Allen's test

INTERVENTIONS:
Other: Allen's test — The Allen's test checks to make sure that radial and ulnar arteries that supply blood to the hand are not blocked. A pulse oximeter is placed on the index finger of the hand. The subject is asked to make a fist for 10 seconds.At this time, pressure is applied over the ulnar and radial arteries as to occlude (block) both of them. The pulse oximeter reading will begin to fall. Radial arterial pressure is then released. If the artery is patent (working), the pulse oximeter reading will begin to rise.
  Groups: Radial
Other: Distal pulses — Practitioner will check that the dorsalis pedis and posterior tibialis are palpable.
  Groups: Femoral

SUMMARY:
Cardiac catheterization has traditionally been performed via access to the arterial circulation from the femoral artery located in the groin. As an alternative to this approach, the radial artery, located in the arm, is gaining wider use in clinical practice. Multiple studies have demonstrated that cardiac catheterization via the radial approach has a very low complication rate, in the short term. This study is intended to determine if there are any differences in the long term complication rate between radial artery cardiac catheterization as compared with femoral artery cardiac catheterization.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* 19 years old or older
* candidate for radial or femoral cardiac catheterization

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting at Creighton University Medical Center Cardiac Catheterization laboratory for either radial or femoral cardiac catherization
Sampling Method: Non-Probability Sample
Enrollment: 243 (Actual)
Dates: Start 2010-06; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
To determine if there is a difference in complication rate measured at 30 days between radial and femoral catheterization | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Michael White, MD, Principal Investigator — Creighton University
Locations (2):
- United States (2):
  - Creighton University Medical Center, Omaha, Nebraska
  - The Cardiac Center at Creighton University, Omaha, Nebraska